CLINICAL TRIAL: NCT03908268
Title: Group Family Nurture Intervention: Short and Long Term Effects on Preschool Aged Children and Their Mothers at Children's Learning Centers
Brief Title: Children's Learning Centers Group FNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Children's Learning Centers of Fairfield County (Unknown)
Responsible Party: Principal Investigator, Martha G Welch, Associate Professor of Psychiatry (in Pediatrics and Pathology and Cell Biology), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AAAS1630
Record Dates: First submitted 2018-12-17; First posted 2019-04-09 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Relation, Mother-Child; Family Conflict; Emotional Disturbances; Behavior Problem; Development Delay
Keywords: Co-regulation; Emotional Connection; Family Nurture Intervention; Preschool Intervention; Martha G. Welch MD; Multiple Family Group Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Affective Symptoms; Mental Disorders; Learning Disabilities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLC Program (Active Comparator): Half of the mother-child dyads who are enrolled in the study will be randomly assigned to the Standard Children's Learning Center Program group.
  Interventions: Behavioral: Standard Children's Learning Center (CLC) Program
- FNI plus CLC Program (Experimental): Half of the mother-child dyads who are enrolled in the study will be randomly assigned to the Family Nurture Intervention plus Standard CLC Program group.
  Interventions: Behavioral: Family Nurture Intervention (FNI)

INTERVENTIONS:
Behavioral: Family Nurture Intervention (FNI) — The mother-child pair will be asked to talk and play with each other as the pair customarily does. If the child becomes restless and dysregulated, the mother will be coached by the Nurture Specialist to bring the child back into a calm state through sustained physical contact, comforting touch, soothing words and eye contact. Each dyad will attend eight group FNI sessions within sixteen weeks.
  Other Names: FNI
  Arms: FNI plus CLC Program
Behavioral: Standard Children's Learning Center (CLC) Program — Typical, age-tailored CLC curriculum taught by CLC teachers. Children attend CLC as usual and parents do not take part in group sessions.
  Other Names: CLC
  Arms: CLC Program

SUMMARY:
The purpose of this study is to compare the effects of Family Nurture Intervention in a mother-child group setting with a Standard Children's Learning Center (CLC) Program for preschool-aged children (ages 2-4.5). This approach is based on creating emotional connection and establishing mother-child two-way regulation, which the investigators hypothesize affects early child development. Mothers and children will be engaged by Nurture Specialists in comforting and calming interactions to regulate each other physically-leading to an automatic calming response to contact with each other.

DETAILED DESCRIPTION:
This study tests a group model of Family Nurture Intervention (FNI), a novel family-based intervention that facilitates mother-child emotional connectedness and co-regulation. Many current interventions aim at helping the child to self-regulate with or without the mother's help. However, according to the investigators' Calming Cycle Theory, the ability of the mother-child dyad to promote optimal development is dependent on the dyad's ability to co-regulate. The interactive co-regulation between the mother and the child shapes the behavior of both. This study aims to investigate the short and long term effects of FNI in a multiple family group setting for preschool aged children to prevent and/or treat developmental/behavioral problems.

Previously, FNI implemented in the Neonatal Intensive Care Unit (NICU) for premature infants and their mothers at Columbia University Medical Center demonstrated that FNI positively alters neurodevelopment of premature infants. Infants who received FNI in the NICU demonstrated increased brain activity in the prefrontal cortex at term age, improved cognitive and language development at 18 months as measured by the Bayley Scales of Infant Development, improved behavior on the Child Behavior Checklist (CBCL) and reduced risk for autism as indicated by the Modified Checklist for Autism in Toddlers (M-CHAT) at 18 months. The pilot study of FNI with preschool aged children and their mothers shows a 40% reduction in behavioral problems on the CBCL. Accordingly, the investigators hypothesize that the Family Nurture Intervention will alter physiological regulatory capacities and will result in improved indices of mother-child emotional connection and other outcomes in the preschool population similar to the results in the preterm population.

ELIGIBILITY:
Inclusion Criteria:

* Mother is able to consent in English or Spanish
* Mother is 18 years of age or older at the time of consent
* Child is between the ages of 2 to 4 years and 9 months at date of enrollment
* Child resides with mother

Exclusion Criteria:

* The child has severe congenital anomalies or chromosomal anomalies including Downs syndrome and Cerebral Palsy
* The child has a diagnosis of Autism Spectrum Disorder
* The child has severe motor or physical disability
* Mother currently presents with psychosis or is currently taking antipsychotic medication
* Current maternal drug and/or alcohol abuse
* Mother is more than four months pregnant
* Mother and/or infant has a medical condition or contagion that precludes intervention components
* Mother is unable to commit to study schedule
* Mother is currently involved with the Department of Children and Families (DCF)

Ages: 24 Months to 57 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Change in Videotaped Interrupted Welch Lap Test | Baseline, after 8 sessions/weeks and at 6-months post-accrual
  Mother-child interactions will be assessed for social engagement and emotional connection via the Welch Emotional Connection Screen (WECS).
  The Welch Emotional Connection Scale (WECS) construct is emotional connection between mother and child, which the investigators hypothesize predicts optimal development. There are four items on the WECS: Mutual Attraction, Mutual Vocal Exchange, Mutual Facial Engagement, and Mutual Sensitivity/Reciprocity. Each item is rated on a scale from 1 to 3 in 0.25 increments with a score of 3 considered optimal. There is also a binary question to the rater asking if the pair is emotionally connected - yes or no. The mother and child are scored as a pair, not individually.

SECONDARY OUTCOMES:
Respiration | Baseline, after 8 sessions/weeks and at 6-months post-accrual
  Using a Biopac respiration belt, the respiration rate of mother and child will be measured during each assessment and used to compute vagal tone.
ECG | Baseline, after 8 sessions/weeks and at 6-months post-accrual
  Using a Biopac heart rate monitor and electrodes, the heart rate of mother and child during assessment will be measured. The change in R-R wave interval of mother and child throughout the assessment will be computed and used to compute vagal tone.
Change in Maternal Symptoms of Anxiety and Depression | Baseline, after 8 sessions/weeks and at 6-months post-accrual
  Measured via self-report on the Center for Epidemiologic Studies Depression Scale (CES-D), which measures symptoms of depression in nine different groups as defined by the American Psychiatric Association Diagnostic and Statistical Manual - Fifth Edition (DSM-V). Mothers are asked to respond to questions such as "I felt hopeful about the future." Responses range from "rarely or none of the time" to "most or all of the time." "Rarely..." earns a 0 while "most..." earns a 3, with the two responses in the middle earning a 1 and a 2. Each item in the CES-D is weighted equally. Scores are summed to equal a total score. A lower total score indicates the individual is minimally depressed (better outcome), whereas a higher total score indicates the individual is more severely depressed (worse outcome).
Change in Maternal Symptoms of Anxiety and Depression | Baseline, after 8 sessions/weeks and at 6-months post-accrual
  Measured via self-report on the Resilience/Stress (R/S) Questionnaire, a metric of the stress and resilience the mother experienced and developed during her childhood. The R/S Questionnaire is presented in a Likert scale format, asking the mother to respond to statements such as "I believe that my mother loved me when I was little." Potential answers range from "definitely true" to "definitely not true," where "definitely true" earns 1 point while "definitely not true" earns 5. Total scores are calculated by summing the points attributed to each response. A lower total score indicates that the mother had a healthy support system and experienced situations benefiting her psychological health. In contrast, multiple statements answered "definitely not true" or "probably not true," indicates a worse outcome, a lack of social support or psychological well-being during the mother's childhood.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Welch, MD, Principal Investigator — Columbia University
Locations (1):
- Children's Learning Centers of Fairfield County, Cos Cob, Connecticut, United States

REFERENCES:
- [Background] Welch MG, Myers MM, Grieve PG, Isler JR, Fifer WP, Sahni R, Hofer MA, Austin J, Ludwig RJ, Stark RI; FNI Trial Group. Electroencephalographic activity of preterm infants is increased by Family Nurture Intervention: a randomized controlled trial in the NICU. Clin Neurophysiol. 2014 Apr;125(4):675-684. doi: 10.1016/j.clinph.2013.08.021. Epub 2013 Oct 17. PMID 24140072
- [Background] Welch MG, Firestein MR, Austin J, Hane AA, Stark RI, Hofer MA, Garland M, Glickstein SB, Brunelli SA, Ludwig RJ, Myers MM. Family Nurture Intervention in the Neonatal Intensive Care Unit improves social-relatedness, attention, and neurodevelopment of preterm infants at 18 months in a randomized controlled trial. J Child Psychol Psychiatry. 2015 Nov;56(11):1202-11. doi: 10.1111/jcpp.12405. Epub 2015 Mar 11. PMID 25763525
- [Background] Myers MM, Grieve PG, Stark RI, Isler JR, Hofer MA, Yang J, Ludwig RJ, Welch MG. Family Nurture Intervention in preterm infants alters frontal cortical functional connectivity assessed by EEG coherence. Acta Paediatr. 2015 Jul;104(7):670-7. doi: 10.1111/apa.13007. Epub 2015 Apr 13. PMID 25772627
- [Derived] Markowitz ES, Maier MC, Ludwig RJ, Austin J, Maybach AM, Jaffe ME, Welch MG. Qualitative insights from a randomized clinical trial of a mother-child emotional preparation program for preschool-aged children. BMC Psychol. 2023 Sep 1;11(1):257. doi: 10.1186/s40359-023-01288-y. PMID 37653536